CLINICAL TRIAL: NCT06272045
Title: Early Intervention to Promote Cardiovascular Health of Mothers and Children (ENRICH)
Brief Title: Early Intervention to Promote Cardiovascular Health of Mothers and Children
Acronym: ENRICH
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: JHSPH Center for Clinical Trials (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: IRB00398712; 5U24HL163114 (NIH)
Record Dates: First submitted 2024-02-15; First posted 2024-02-22 (Actual); Last update posted 2025-10-20 (Actual); Status verified 2025-10

CONDITIONS: Cardiovascular Health
Keywords: Home visiting, cardiovascular health, prevention, maternal-child health

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: cluster randomized at the home visiting supervisor level, stratified within home visiting agencies
  Participants are masked throughout the study enrollment process (e.g., recruitment, consent, and baseline data collection). Participant may become unmasked to treatment arm after enrollment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ENRICHed home visiting (Experimental): Home Visiting with the addition of cardiovascular health promotion content
  Interventions: Behavioral: ENRICH
- Usual Home Visiting (Active Comparator): Usual home visiting without cardiovascular health promotion content
  Interventions: Behavioral: Usual Home Visiting

INTERVENTIONS:
Behavioral: ENRICH — In the ENRICH intervention, home visitors will incorporate heart health information and activities into routine home visits beginning in pregnancy and continuing until children turn 2 years old. The intervention includes 1) Information and resources on topics such as healthy eating, physical activity, weight management, tobacco use, healthy sleep and stress reduction, 2) tools like scales, Fitbits, and blood pressure monitors to facilitate self-monitoring, and 3) activities and information focused on infant nutrition, feeding, healthy growth, sleep, play and emotions and soothing.
  Arms: ENRICHed home visiting
Behavioral: Usual Home Visiting — Usual home visiting without cardiovascular health promotion content
  Arms: Usual Home Visiting

SUMMARY:
Early Intervention to Promote Cardiovascular Health of Mothers and Children (ENRICH) is a cluster randomized clinical trial, funded by the National Heart Lung & Blood Institute. The study is designed to test the effectiveness of home visiting intervention to promote cardiovascular health and reduce disparities in maternal and early childhood cardiovascular health. Sites, in partnership with evidence-based home visiting programs, are recruiting 6618 participants in total (i.e., 3309 mother-child dyads which includes 3309 mothers and 3309 children) from diverse community settings with a high burden of cardiovascular disease risk factors.

ELIGIBILITY:
Inclusion Criteria:

1. Be currently enrolled in an evidence-based home visiting program participating in ENRICH
2. Be pregnant, with a single or multifetal gestation, at or less than 34 weeks 0 days gestation (per self-report at time of consent)
3. Be 18 years of age or older
4. Speak English or Spanish

Exclusion Criteria: There are no exclusion criteria being applied in assessing eligibility for participation in ENRICH.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 6618 (Estimated)
Dates: Start 2024-06-19 (Actual); Primary Completion 2027-09 (Estimated); Study Completion 2028-07 (Estimated)

PRIMARY OUTCOMES:
Parent physical activity | 12 months after birth
  Time spent in moderate and vigorous physical activity in parent participants
Parent diet measured by Mediterranean Eating Pattern for Americans (MEPA) scale | 12 months after birth
  Diet quality among parent participants as measured by Mediterranean Eating Pattern for Americans (MEPA) scale. The MEPA is a 16-item dietary screener designed to assess accordance with the Mediterranean-like diet patterns during the past 7 days among adults. A score of '0' will be given if the scoring condition is not met and a score of '1' will be given if the scoring condition is met. A score of '1' for any given item was indicative of Mediterranean-like diet accordance. If any condition was not met, a score of '0' was recorded for that item. The total MEPA score could range from 0 to 16. Scores will be converted to points on a 100-point scale based on quantiles of the 16-item measure. For example, scores from 0-3 (0 points), 4-7 (25 points), 8-11 (50 points), 12-14 (80 points), and 15-16 (100 points). Higher scores mean that the adult's diet is similar to a Mediterranean diet.
Parent body mass index | 12 months after birth
  Body mass index (BMI) of parent participants
Parent blood pressure | 12 months after birth
  blood pressure (BP) in parent participants

SECONDARY OUTCOMES:
Child body mass index | 24 months old
  body mass index in child

CONTACTS AND LOCATIONS:
Locations (9):
- United States (9):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - California Polytechnic State University, San Luis Obispo, California
  - University of Colorado, Aurora, Colorado
  - Northwestern University, Chicago, Illinois
  - Washington University in St. Louis, St Louis, Missouri
  - Wake Forest University, Winston-Salem, North Carolina
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - Pennsylvania State University, State College, Pennsylvania
  - Brown University/Lifespan, Providence, Rhode Island

IPD SHARING:
Plan to Share IPD: No